CLINICAL TRIAL: NCT05079932
Title: Pilot Study for the Evaluation of Food Choices and Exclusion of Gluten From the Diet in Patients With Inflammatory Bowel Diseases
Brief Title: Pilot Study for the Evaluation of Food Choices in Patients With Inflammatory Bowel Diseases (MICI2021)
Acronym: MICI2021
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Luca Elli, MD, PhD, Principal Investigator, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Other Study IDs: 612_2021
Record Dates: First submitted 2021-09-23; First posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Ulcerative rectocolitis; Crohn Disease; Gluten-free diet; IBD; Nutrition
MeSH Terms: conditions — Inflammatory Bowel Diseases; Proctocolitis; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project is a pilot study exploring the effects of dietary choices and quantitative digestion of gluten ingested by individuals with IBD compared to a control population. The aim of the study is to evaluate for the first time in an Italian population of subjects with IBD the presence of a diet based on GFD (gluten free diet).

DETAILED DESCRIPTION:
Subjects with IBD will be recruited among the patients referred to the IBD clinic of the Policlinico of Milan. These patients are subject to annual check-ups during which, where possible, they will be asked to sign an informed consent. These patients are subjected during the visits of normal clinical follow-up to:

* Questionnaire on eating habits for the patient with IBD versus control patients;
* Modified Food Habits Frequency Questionnaire (FFQ), validated for the celiac population. The questionnaire assesses the extent, frequencies of consumption and quantity of gluten-containing foods in a year; this, in order to estimate the average introduction of gluten through the diet versus control patients;
* Anthropometric and plicometric analysis;
* Validated clinical activity questionnaires for RCU (ulcerative rectocolitis) and CD (Chron disease) (Mayo Score and Harvey-Bradshaw Index).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years
* Gender: women and men
* Patients who have been diagnosed with IBD for at least 12 months
* patients who have signed an informed consent

Exclusion Criteria:

* Pregnancy status
* Patients not suffering from the two main forms of IBD, i.e. CD or RCU (unclassified IBD colitis, collagenous colitis, lymphocytic colitis will be excluded).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 patients with IBD (15 CD and 15 RCU) and 15 patients from the control population
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Dietary habits in IBD patients | April 2021- April 2023
  Quantification of gluten intake by IBD patients compared with the control population.
  Evaluation of foods excluded from the diet of IBD patients.

SECONDARY OUTCOMES:
Assessment of weight | April 2021- April 2023
  Assessment of weight (kilograms) in IBD patients
Assessment of height | April 2021- April 2023
  Assessment of height (meters) in IBD patients
Assessment of clinical disease activity | April 2021- April 2023
  Evaluation of validated clinical activity indices for RCU in IBD patients (Mayo Score)
Assessment of clinical disease activity | April 2021- April 2023
  Evaluation of validated clinical activity indices for CD in IBD patients (Harvey-Bradshaw Index)

CONTACTS AND LOCATIONS:
Overall Officials: Luca Elli, PhD, Principal Investigator — Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano, Milan, Italy

REFERENCES:
- [Result] Weaver KN, Herfarth H. Gluten-Free Diet in IBD: Time for a Recommendation? Mol Nutr Food Res. 2021 Mar;65(5):e1901274. doi: 10.1002/mnfr.201901274. Epub 2020 Jun 28. PMID 32558265
- [Result] Mazzeo T, Roncoroni L, Lombardo V, Tomba C, Elli L, Sieri S, Grioni S, Bardella MT, Agostoni C, Doneda L, Brighenti F, Pellegrini N. Evaluation of a Modified Italian European Prospective Investigation into Cancer and Nutrition Food Frequency Questionnaire for Individuals with Celiac Disease. J Acad Nutr Diet. 2016 Nov;116(11):1810-1816. doi: 10.1016/j.jand.2016.04.013. Epub 2016 May 28. PMID 27245762
- [Result] Schroeder KW, Tremaine WJ, Ilstrup DM. Coated oral 5-aminosalicylic acid therapy for mildly to moderately active ulcerative colitis. A randomized study. N Engl J Med. 1987 Dec 24;317(26):1625-9. doi: 10.1056/NEJM198712243172603. PMID 3317057
- [Result] Dhanda AD, Creed TJ, Greenwood R, Sands BE, Probert CS. Can endoscopy be avoided in the assessment of ulcerative colitis in clinical trials? Inflamm Bowel Dis. 2012 Nov;18(11):2056-62. doi: 10.1002/ibd.22879. Epub 2012 Jan 23. PMID 22271464
- [Result] Harvey RF, Bradshaw JM. A simple index of Crohn's-disease activity. Lancet. 1980 Mar 8;1(8167):514. doi: 10.1016/s0140-6736(80)92767-1. No abstract available. PMID 6102236
- [Result] Elli L, Bascunan K, di Lernia L, Bardella MT, Doneda L, Soldati L, Orlando S, Ferretti F, Lombardo V, Barigelletti G, Scricciolo A, Fabiano S, Vecchi M, Roncoroni L. Safety of occasional ingestion of gluten in patients with celiac disease: a real-life study. BMC Med. 2020 Mar 16;18(1):42. doi: 10.1186/s12916-020-1511-6. PMID 32172690